CLINICAL TRIAL: NCT03326349
Title: Home-based Computerized Cognitive Rehabilitation in Chronic Stage Stroke
Acronym: CHRONIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josep M. Tormos Muñoz (Other)
Responsible Party: Sponsor-Investigator, Josep M. Tormos Muñoz, Research Director, Institut Guttmann
Organization: Institut Guttmann (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2016251
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Chronic Stroke; Cognitive Impairment
Keywords: computerized cognitive rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guttmann, NeuroPersonalTrainer (Experimental): Guttmann NeuroPersonalTrainer (GNPT) 5 days per week over 6 weeks.
  Interventions: Other: Guttmann, NeuroPersonalTrainer
- Ictus.online (Sham Comparator): Itus.online 5 days per week over 6 weeks
  Interventions: Other: Ictus.online

INTERVENTIONS:
Other: Guttmann, NeuroPersonalTrainer — Guttmann NeuroPersonalTrainer (GNPT) is a telerehabilitation platform. GNPT consists of a set of computerized cognitive exercises covering different cognitive functions and subfunctions. Every task has been specifically based on cognitive paradigms to address specific cognitive subfunction. The rehabilitation process starts by assigning a patient to a therapist responsible for the treatment. The therapist has then to perform the initial neuropsychological assessment, consisting of a set of validated tests used to attention, memory and executive functions prior to the treatment. The results of these tests will be stored in GNPT system. Then, the cognitive profile is calculated using these results, and taking into account the patient's age and study level. Using this profile, the program assigns a set of computerized tasks to a certain day, configuring the input parameters of each task in order to personalize treatments.
  Arms: Guttmann, NeuroPersonalTrainer
Other: Ictus.online — An online domain which provides a daily session of one hour of duration. Each session consists of four ten-minute videos. After each video, the participant must complete a three-question quiz about the contents of the video (for example, "What animal appears in in the video?"). The difficulty level is minimal, and does not vary depending on the execution of the participant.
  Arms: Ictus.online

SUMMARY:
This study evaluates the effectiveness of Guttmann NeuroPersonalTrainer (GNPT), a tele-rehabilitation platform developed as a tool for the cognitive rehabilitation of chronic stroke patients. All patients will receive this treatment but in different order: half will receive GNPT and the other half will receive sham cognitive training; after a washout period of three months, crossover will occur and participants from the GNPT condition will receive sham cognitive training, while participants originally from the control intervention will receive GNPT.

ELIGIBILITY:
Inclusion Criteria:

* to be over 18 years old,
* to have been diagnosed with stroke
* an occurrence of the injury of 12 month period ore more (chronic stage)
* cognitive impairment confirmed by pre-intervention neuropsychological assessment

Exclusion Criteria:

* diagnosis of language deficits or aphasia
* motor impairment concerning upper limbs that may incapacitate them for the use of the computer
* severe alteration of the visual field or perceptual problems
* health status that may require further intervention or admission to a medical center during the study;
* neurological or psychiatric history
* substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Conners Continuous Performance Test (CPT-II) | 1 day
  To improve performance in sustained attention after receiving experimental intervention.
Rey Auditory Verbal Learning Test (RAVLT) | 1 day
  To improve performance in short-term, long-term and recognition. This test has puntuation range from 0 to 75.
Spanish phonemic fluency test- PMR | 1 day
  To improve performance in phonemic fluency after receiving experimental intervention.
Digit Span forward Subtest from the Wechsler Adult Intelligence Scale (WAIS-III) | 1 day
  To improve performance in span of immediate verbal recall after receiving experimental intervention. This subtest has a puntuation range from 2 to 9, where higher values are considered to be a better outcome.
Digit Span backward Subtest from the Wechsler Adult Intelligence Scale (WAIS-III) | 1 day
  To improve performance in working memory after receiving experimental intervention. This subtest has a puntuation range from 2 to 8, where higher values are considered to be a better outcome.
Letter-Number Sequencing Subtest from the Wechsler Adult Intelligence Scale (WAIS-III) | 1 day
  To improve performance in working memory after receiving experimental intervention. This subtest has a puntation range from 1 to 21, where higher values are considered to be a better outcome.
Rating Scale for Attentional Behavior (RSAB) | 1 week
  RSAB comprises 14 items aimed to identify attentional difficulties on daily routines
Prospective and Retrospective Memory Questionnaire (PRMQ) | 1 week
  PRMQ includes 16 items designed to evaluate prospective and retrospective memory in short- and long-term
Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) | 1 week
  BRIEF-A includes 75 items designed to assess executive function behaviors on day-to-day activities.

SECONDARY OUTCOMES:
Digit Symbol-Coding Subtest from the Wechsler Adult Intelligence Scale (WAIS-III) | 1 day
  To improve performance in speed of processing. This subtest has a puntuation range from 1 to 133, where higher values are considered to be a better outcome.
Block Design Subtest from the Wechsler Adult Intelligence Scale (WAIS-III) | 1 day
  To improve performance in visuoconstruction and planning. This subtest has a puntuation range from 1 to 68, where higher values are considered to be a better outcome.
Stroop Color and Word test (Stroop Test) | 1 day
  To improve performance in inhibitory control
Trail Making Test A (TMT-A) | 1 day
  To improve performance in visual attention
Trail Making Test B (TMT-B) | 1 day
  To improve performance in task-switching
Wisconsin Card Sorting Test (WCST) | 1day
  To improve performance in cognitive flexibility

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Guttmann, Barcelona, Spain

REFERENCES:
- [Derived] Gibson E, Koh CL, Eames S, Bennett S, Scott AM, Hoffmann TC. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD006430. doi: 10.1002/14651858.CD006430.pub3. PMID 35349186
- [Derived] Gil-Pages M, Solana J, Sanchez-Carrion R, Tormos JM, Ensenat-Cantallops A, Garcia-Molina A. A customized home-based computerized cognitive rehabilitation platform for patients with chronic-stage stroke: study protocol for a randomized controlled trial. Trials. 2018 Mar 22;19(1):191. doi: 10.1186/s13063-018-2577-8. PMID 29566766